CLINICAL TRIAL: NCT02046460
Title: Biomarkers and Antithrombotic Treatment in Cervical Artery Dissection - TREAT-CAD
Acronym: TREAT-CAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stefan Engelter (Other)
Responsible Party: Sponsor-Investigator, Stefan Engelter, Prof. Dr. med., MD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 340/12
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Cervical Artery Dissection
MeSH Terms: interventions — Aspirin; acarboxyprothrombin; Phenprocoumon; Warfarin; Acenocoumarol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: PROBE-Design: Prospective, randomized, open-label, blinded assessment of end-points.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Anticoagulation (Active Comparator): Vitamin K-Antagonists, target INR 2.0-3.0
  Interventions: Drug: Vitamin K antagonist
- Antiplatelets (Experimental): Acetylsalicylic acid, 300mg o.p.d.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Acetylsalicylic acid — Acetylsalicylic acid, 300mg o.p.d.
  Other Names: ASA
  Arms: Antiplatelets
Drug: Vitamin K antagonist — Vitamin K-antagonists, target INR 2.0-3.0
  Other Names: Phenprocoumon, Warfarin, Acenocoumarol
  Arms: Oral Anticoagulation

SUMMARY:
Primary objective: To demonstrate the non-inferiority of acetylsalicylic acid (ASA) to anticoagulant treatment (vitamin K antagonists) in CAD-patients with regard to outcome and complication measures.

Methods: Randomized controlled, open labeled multicenter, non-inferiority trial with blinded assessment of outcome events.

Primary endpoint: Primary composite outcome measure - labeled Cerebrovascular Ischemia, major Hemorrhagic events or Death (CIHD) - includes the following efficacy and safety outcome measures during the treatment period: (i) occurrence of any stroke*, new acute lesions on diffusion weighted MRI (ii) any major extracranial hemorrhage, any symptomatic intracranial hemorrhage and any asymptomatic micro- or macrobleeds, (iii) death.

DETAILED DESCRIPTION:
Substudies:

1. In-depth analysis of the TREAT-CAD randomized trial:

   The investigators will perform a subgroup analysis on the per-protocol population investigating if the antithrombotic treatment effect (anticoagulation versus aspirin) depends on specific patient baseline characteristics. The investigators will look at the following subgroups: Presenting with cerebral ischemia - either clinical ischemic events, MRI lesions, or both - versus presenting with local symptoms only, occlusion of the dissected artery at baseline (no/yes), early versus delayed treatment start (divided by the median of the study population), acute recanalization therapy including intravenous thrombolysis and/or endovascular therapy (no/yes), intracranial extension of the dissected artery (no/yes), site of dissection defined as internal carotid artery dissection versus vertebral artery dissection, single versus multivessel dissection, younger versus older age (divided by the median of the study population), and male versus female.
2. TCD Monitoring Substudy:

   The objective of the TREAT-CAD transcranial Doppler (TCD) substudy is to (i) detect the frequency of microembolic signals (MES) in CAD patients, stratified to the type of treatment (aspirin vs. anticoagulation) - in the setting of an RCT (randomized controlled trial)- and (ii) to evaluate the meaning of MES by addressing the following questions: (a) Is there an association of MES (presence or number) with the occurrence of clinical and/or surrogate MR (magnetic resonance) outcome measures; (b) Is there an interaction between MES, type of treatment and outcome events. Participants are asked to allow a 6-h TCD monitoring in between day 1 and day 4 since start of the allocated study treatment. Recordings were allowed to be split in up to three episodes (2 h each). In patients with ICAD (internal carotid artery dissection), the ipsilateral middle cerebral artery is investigated. In patients with VAD (vertebral artery dissection), the ipsilateral posterior cerebral artery is investigated.
3. Biomarker substudy:

   The objective of the biomarker study is to investigate whether the plasma level of MMP9 (matrix-metalloproteinase 9) and the ratio of the plasma MMP9 to TIMP2 (tissue inhibitor of metalloproteinases 2) is associated with efficacy and safety measures in CAD patients, when stratified to the allocated treatment regime. Plasma samples are collected from participants at baseline (i.e., prior to start of the allocated treatment within the TREAT-CAD main study) and at Follow-up visit 1. The specific focus on MMP9 and TIMP2 is based on preliminary observational data pointing to higher MMP9 and MMP9/TIMP2 ratios in CAD versus control patients.
4. 6 Month-follow-up for TREAT-CAD To compare (i) the frequency of clinical and MRI outcomes 6 months after cervical artery dissection among the per-protocol participants of the TREAT-CAD trial and (ii) to focus on events occurring between 3 and 6 months, stratified to the type of antithrombotic medication taken (as-treated analysis).
5. Detailed imaging analysis in the TREAT-CAD study To identify possible imaging risk factors for recurrent stroke and to evaluate the dependence of antithromobotic therapy on imaging factors.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic or non-ischemic symptoms within 2 weeks
2. Verification of CAD-diagnosis (carotid and/or vertebral) by MR-techniques (at least one):

   * mural hematoma or
   * pseudo-aneurysm or
   * long filiform stenosis or
   * intimal flap or
   * double lumen or
   * occlusion situated more than 2 cm above the bifurcation of the carotid artery, revealing a pseudo aneurysm or a long filiform stenosis after recanalisation.
3. Written informed consent by patient or next-to-kin
4. 24h latency period in case of thrombolysis
5. Age > 18 years by time of inclusion

Exclusion Criteria:

1. MR-contraindications (claustrophobia precluding MRI: patients agreeing to undergo MRI scanning with mild sedation may be entered into the study)
2. Contraindications to the use of anticoagulation (vitamin k antagonists, heparin) or ASA (according to the Swiss "Arzneimittelkompendium" http://www.compendium.ch/search/de or the "Rote Liste" (German centers) or "Lægemiddelstyrelsen - produktresume" for the Danish center (https://laegemiddelstyrelsen.dk/da/bivirkninger/find-medicin/produktresumeer/) and the judgment of the treating physician)
3. Pregnancy (Note: for women in child bearing age a pregnancy test has to be done prior to study entry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Primary composite outcome measure - labeled Cerebrovascular Ischemia, major Hemorrhagic events or Death (CIHD) - | 3 months
  CIHD - includes the following efficacy and safety outcome measures during the treatment period: includes the following efficacy and safety outcome measures during the treatment period: (i) occurrence of any stroke (including retinal infarction), new acute lesions on diffusion weighted MRI (ii) any major extracranial hemorrhage, any symptomatic intracranial hemorrhage and any asymptomatic micro- or macrobleeds, (iii) death.

SECONDARY OUTCOMES:
new ischemic strokes (including retinal infarction) | 3 months
new acute lesions on diffusion-weighted MRI | 3 months
any major extracranial hemorrhage | 3 months
any symptomatic intracranial hemorrhage | 3 months
any asymptomatic micro- or macrobleeds | 3 months
any death | 3 months
any increase in volume of the vessel wall hematoma at the followup cervical MRI as compared to the baseline MR-scan | 3 months
independence in activity of daily living (modified Rankin scale 0-2) at 3 months and at 6 months | 3 months
excellent functional outcome (modified Rankin scale 0,1) at 3 month and at 6 months | 3 months
any TIA (classical definition) | 3 months
recurrent cervical artery dissection | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan T. Engelter, MD, Principal Investigator — University Hospital, Neurorehab. Felix Platter, University of Basel, Switzerland
Locations (10):
- University Hospital, Stroke Center Bispebjerg Hospital Copenhagen, Denmark, Copenhagen, Denmark
- Germany (2):
  - University Hospital, Stroke Center Charite Berlin, Germany, Berlin
  - University Hospital, Stroke Center LMU Munich, Germany, Munich
- Switzerland (7):
  - Kantonsspital, Stroke Center Aarau, Switzerland, Aarau
  - University Hospital, Stroke Center Basel, Switzerland, Basel
  - University Hospital, Stroke Center Inselspital Berne, Switzerland, Bern
  - University Hospital, Stroke Center Geneva, Switzerland, Geneva
  - University Hospital, Stroke Center CHUV Lausanne, Switzerland, Lausanne
  - Kantonsspital, Stroke Center St. Gallen, Switzerland, Sankt Gallen
  - University Hospital, Stroke Center Zurich, Switzerland, Zurich

REFERENCES:
- [Background] Traenka C, Gensicke H, Schaedelin S, Luft A, Arnold M, Michel P, Kagi G, Kahles T, Nolte CH, Kellert L, Rosenbaum S, Sztaizel R, Brehm A, Stippich C, Psychogios M, Lyrer P, Engelter ST; TREAT-CAD investigators. Biomarkers and antithrombotic treatment in cervical artery dissection - Design of the TREAT-CAD randomised trial. Eur Stroke J. 2020 Sep;5(3):309-319. doi: 10.1177/2396987320921151. Epub 2020 Jun 29. PMID 33072885
- [Background] Engelter ST, Traenka C, Gensicke H, Schaedelin SA, Luft AR, Simonetti BG, Fischer U, Michel P, Sirimarco G, Kagi G, Vehoff J, Nedeltchev K, Kahles T, Kellert L, Rosenbaum S, von Rennenberg R, Sztajzel R, Leib SL, Jung S, Gralla J, Bruni N, Seiffge D, Feil K, Polymeris AA, Steiner L, Hamann J, Bonati LH, Brehm A, De Marchis GM, Peters N, Stippich C, Nolte CH, Christensen H, Wegener S, Psychogios MN, Arnold M, Lyrer P; TREAT-CAD investigators. Aspirin versus anticoagulation in cervical artery dissection (TREAT-CAD): an open-label, randomised, non-inferiority trial. Lancet Neurol. 2021 May;20(5):341-350. doi: 10.1016/S1474-4422(21)00044-2. Epub 2021 Mar 23. PMID 33765420
- [Derived] Engelter ST, Enz LS, Ravanelli F, Kaufmann JE, Gensicke H, Schaedelin S, Luft AR, Globas C, Goeggel-Simonetti B, Fischer U, Strambo D, Kagi G, Nedeltchev K, Kahles T, Kellert L, Rosenbaum S, von Rennenberg R, Brehm A, Seiffge D, Renaud S, Brandt T, Sarikaya H, Zietz A, Wischmann J, Polymeris AA, Fischer S, Bonati LH, De Marchis GM, Peters N, Nolte CH, Christensen H, Wegener S, Psychogios MN, Arnold M, Lyrer P, Traenka C. The 6-months follow-up of the TREAT-CAD trial: Aspirin versus anticoagulation for stroke prevention in patients with cervical artery dissection. Eur Stroke J. 2025 Sep;10(3):871-881. doi: 10.1177/23969873251315362. Epub 2025 Feb 5. PMID 39910883

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT02046460/SAP_000.pdf